CLINICAL TRIAL: NCT01997385
Title: The Clinical Effects of Korean Adapted APD in Automated Peritoneal Dialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fresenius Medical Care Korea (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KAAPD_01_112013
Record Dates: First submitted 2013-11-13; First posted 2013-11-28 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Renal Insufficiency, Chronic
Keywords: adapted APD; dwell time; fill volume
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- KAPD-C (Active Comparator): KAPD-C is a treatment prescribed 2000 mL fill volume per each 4 cycles of dialysis session with an exchange cycle of 90 minutes.
  Interventions: Procedure: KAPD-C
- KAPD-A (Experimental): KAPD-A is a treatment initially prescribed 1500 mL fill volume per each 2 cycles of dialysis session with an exchange cycle of 45 minutes and followed by 2 cycles of 2500 mL fill volume with an exchange cycle of 135 minutes.
  Interventions: Procedure: KAPD-A

INTERVENTIONS:
Procedure: KAPD-C — KAPD-C is a treatment prescribed 2000 mL fill volume per each 4 cycles of dialysis session with an exchange cycle of 90 minutes.
  Arms: KAPD-C
Procedure: KAPD-A — KAPD-A is a treatment initially prescribed 1500 mL fill volume per each 2 cycles of dialysis session with an exchange cycle of 45 minutes and followed by 2 cycles of 2500 mL fill volume with an exchange cycle of 135 minutes.
  Arms: KAPD-A

SUMMARY:
The aim of this study is to assess the impact of "adapted" Automated Peritoneal Dialysis(APD) sequentially prescribed shorter and longer dwell exchanges with smaller and larger fill volumes in comparison with "conventional APD" prescribed a standard continuous cycling peritoneal dialysis on the efficacy of dialysis.

DETAILED DESCRIPTION:
It is well known that the efficiency of peritoneal dialysis (PD) varies with the duration of the dwell and the prescribed fill volume. Short dwell ensures adequate UF because the osmotic gradient is maintained while prolonged dwell allows for more solute clearance because the dialysate-to-plasma ratio (D/P) for uremic toxins such as creatinine and phosphate enhances. In terms of intraperitoneal fill volume, large fill volume improves the removal of uremic toxins for two reasons: a larger volume can be drained and therefore the clearance achieved is greater, and the peritoneal surface area available for the exchange is increased. Conversely, small fill volume promotes the process of UF because of the potentially low intraperitoneal pressure (IPP). Overall, choosing the optimal dwell time and exchange volume should promote UF and increase the removal of uremic toxins-urea in particular-to the dialysate.

Thus, this study proposes a new way of giving PD, using a modified version of conventional prescription which firstly uses 2 cycles of short dwell time with a small fill volume to promote UF and subsequently uses 2 cycles of longer dwell time and a larger fill volume to promote removal of uremic toxins from the blood.

Although it was already evaluated the efficiency of this modified prescription by Fischbach et al, the prescription currently prescribed in most Korean hospitals shows some differences in dwell time, fill volume and exchange cycling. The aim of this study is to assess the clinical effect of "Korean Adapted APD" (KAPD-A) compared to "Korean Conventional APD" (KAPD-C).

This is a multicenter, randomized, open-label, parallel controlled study. Patients who meet inclusion criteria will be randomized into each group at the ratio of 1:1. For incident patients, after being stable on APD and peritonitis-free at least 4 weeks, which is called as "run-in period", group 1 will start with 8 weeks of KAPD-C treatment and then cross over to 8 weeks of treatment with KAPD-A while group 2 will be performed on the contrary from KAPD-A to KAPD-C treatment.

Each patient will receive the same total amount of dialysate (8000 mL), given over the same 8-hour duration. First at the inclusion visit called "as baseline", and then visits will take place every 4 weeks for a total of 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* End stage of Renal Disease(ESRD) patients with indication for renal replacement therapy
* D/P Creatinine above 0.5 as evaluated by a 4-hour peritoneal equilibration test(PET) at screening
* Stable on APD and peritonitis-free for at least 4 weeks(run-in phase) in case of incident patients who chose APD
* Peritonitis-free within 4 weeks in case of maintaining patients who treated with APD in current
* Written informed consent to study participation and data submission

Exclusion Criteria:

* Planned to kidney transplantation within 5 months
* Patients with ascites because of the progressed cirrhosis of the liver
* Suspected or confirmed pregnancy
* Prior enrolment in another clinical trial

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1075 (Actual)
Dates: Start 2012-06; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Difference in overnight peritoneal ultrafiltration (UF) between KAPD-C and KAPD-A | at 4,8,12,16 weeks from baseline
Difference in weekly peritoneal Kt/V urea between KAPD-C and KAPD-A | at 4,8,12,16 weeks from baseline
Difference in weekly peritoneal creatinine clearance between KAPD-C and KAPD-A | at 4,8,12,16 weeks from baseline

SECONDARY OUTCOMES:
Difference in phosphate dialytic removal between KAPD-C and KAPD-A | at 4,8,12,16 weeks from baseline
Difference in corrected for glucose absorption between KAPD-C and KAPD-A | at 4,8,12,16 weeks from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Daejoong Kim, Prof., Principal Investigator — Division of Nephrology, Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No